CLINICAL TRIAL: NCT02157571
Title: A Multi-center, Randomized, Double-blind, Double-dummy Clinical Study to Evaluate the Safety and Efficacy of Prulifloxacin Film-coated Tablet for the Treatment of Acute Exacerbations of Chronic Bronchitis With Levofloxacin Hydrochloride Tablet as Active Control
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prulifloxacin AECB ZK-004
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Acute Exacerbations of Chronic Bronchitis
Keywords: prulifloxacin; AECB; Levofloxacin
MeSH Terms: interventions — prulifloxacin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prulifloxacin (Experimental): Prulifloxacin film-coated tablet : 600 mg/tablet, oral administration of a single tablet.
  Placebo of levofloxacin hydrochloride tablet, without active components.
  Interventions: Drug: Prulifloxacin; Drug: Levofloxacin Placebo
- Levofloxacin (Active Comparator): Levofloxacin hydrochloride tablet 500 mg/tablet, oral administration of a tablet daily.
  Placebo of prulifloxacin film-coated tablet without active components.
  Interventions: Drug: Levofloxacin; Drug: Prulifloxacin placebo

INTERVENTIONS:
Drug: Prulifloxacin — 600 mg/tablet, oral administration of a single tablet.
  Arms: Prulifloxacin
Drug: Levofloxacin — 500 mg/tablet, oral administration of a tablet daily.
  Arms: Levofloxacin
Drug: Levofloxacin Placebo — Placebo of levofloxacin hydrochloride tablet, without active components.
  Arms: Prulifloxacin
Drug: Prulifloxacin placebo — Placebo of prulifloxacin film-coated tablet without active components.
  Arms: Levofloxacin

SUMMARY:
The purpose of this study is to use oral prulifloxacin to treat patient with Acute Exacerbations of Chronic Bronchitis and compare the effect with Levofloxacin.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing to participate in the study and gives the signature of informed consent;
2. In and out-patients (aged 18-70 years old), male or female;
3. Patient receives no effective antibacterial therapy or the therapy has no remarkable efficacy, or positive bacterial test result in the past 72 hours;
4. Diagnosed as mild to moderate acute exacerbation of chronic bronchitis patients (see <Severity Evaluation Criteria Table>)
5. Within 48 hours prior to the study, women of child-bearing age have a negative urine pregnancy test and is willing to use efficient measures of contraception to avoid pregnancy during the study.

Exclusion Criteria:

1. Patient hypersensitive to quinolones or with allergic constitution;
2. Patient with severe condition which need combination with other antibacterial agents;
3. Concurrent infections in other organs or system;
4. Patient with severe heart, liver or kidney disease, or Q-T prolongation of over 450 ms, serum AST or ALT more than twice as high as the upper limit of normal or Cr over the upper limit of normal;
5. With any of the following diseases: active tuberculosis, bronchiectasis, lung abscess, aspiration pneumonia, lung cancer, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pulmonary embolism, pulmonary addicted acidic granulocyte infiltration and pulmonary vasculitis syndrome;
6. Patient with severe hematologic disease or central nervous system disease or convulsion history, with mental status unable to coordinate;
7. Patient with malignant tumor or other severe background disease;
8. Patient with severe immunodeficiency;
9. A history of tendon;
10. Known pregnancy or lactation;
11. Prulifloxacin contains lactose, therefore, patients with a rare genetic disease such as galactose intolerance, Lapp lactase deficiency or glucose - galactose malabsorption cannot be enrolled;
12. Participation in other clinical trials within 3 months before screening or currently on any investigational therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of prulifloxacin film-coated tablet in the treatment of acute exacerbations of chronic bronchitis. | 7-10 days
  1. Clinical efficacy: consists of clinical evaluation which expressed as clinical cure and clinical failure.
  2. Bacteriological efficacy: consists of eradication, supposed eradication, persistence, supposed persistence, partial eradication,;
  3. Comprehensive therapeutic efficacy: consists of cure and failure

SECONDARY OUTCOMES:
safety of treatment | 7-10 days
  Vital signs, ECG, laboratory examinations and adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Nei Mongo medical University, Nei Mongo, China